CLINICAL TRIAL: NCT02038010
Title: A Phase I Study of BYL719 and Trastuzumab-MCC-DM1 in HER2-Positive Metastatic Breast Cancer Patients With Progression on Prior Trastuzumab and Taxane-Based Therapy
Brief Title: BYL719 + T-DM1 in HER2(+) Metastatic Breast Cancer Pts Who Progress on Prior Trastuzumab & Taxane Tx
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Novartis (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Gradishar, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 13B06; NCI-2013-02224 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NU 13B06 (Other: Northwestern University); P30CA060553 (NIH); STU00087202 (Other: Northwestern University IRB#)
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: HER2-positive Breast Cancer; Recurrent Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Alpelisib; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (PI3K inhibitor BYL719, ado-trastuzumab emtansine) (Experimental): Patients receive PI3K inhibitor BYL719 PO daily on days 1-21 and ado-trastuzumab emtansine IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PI3K inhibitor BYL719; Biological: ado-trastuzumab emtansine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: PI3K inhibitor BYL719 — Given PO
  Other Names: BYL719; phosphoinositide 3-kinase inhibitor BYL719
Biological: ado-trastuzumab emtansine — Given IV
  Other Names: Kadcyla; T-DM1; trastuzumab-DM1; trastuzumab-MCC-DM1; trastuzumab-MCC-DM1 antibody-drug conjugate
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
The purpose of this study is to see whether a combination of two different drugs - trastuzumab-MCC-DM1 (T-DM1) and BYL719 is safe, and if it might be effective in treating metastatic breast cancer. T-DM1 is a type of drug that contains an antibody (trastuzumab) linked to chemotherapy. The antibody in T-DM1 targets a marker on breast cancer cells called HER2, which allows the drug to go directly to the cancer cells. The use of T-DM1 in this study is considered standard treatment for the type of cancer in this study. Participants in this study have already been treated with trastuzumab and chemotherapy in the past, and their cancer has gotten worse in spite of those treatments. BYL719 is an oral drug (taken by mouth) that the researchers think may help T-DM1 to work better.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine safety, tolerability, feasibility, and the maximum-tolerated dose (MTD) of dose-escalating BYL719 in combination with ado-trastuzumab emtansine (T-DM1) in patients with HER2-positive metastatic breast cancer (MBC) after progression on trastuzumab and taxane-based therapy.

SECONDARY OBJECTIVES:

I. Evaluate pharmacokinetics (PK) of BYL719 administered in combination with T-DM1.

II. Assess any preliminary evidence of efficacy of BYL719 and T-DM1 in combination in patients with HER2-positive MBC.

TERTIARY OBJECTIVES:

I. Explore efficacy in patients whose tumors have an alteration (mutation or amplification) of the PIK3CA gene and decrease of phosphatase and tensin homolog gene (PTEN) expression. (Optional) II. Examine other v-akt murine thymoma viral oncogene homolog 1 (Akt)/mechanistic target of rapamycin (mTOR) downstream markers by immunohistochemistry. (Optional)

OUTLINE: This is a dose-escalation study of PI3K inhibitor BYL719.

Patients receive PI3K inhibitor BYL719 orally (PO) daily on days 1-21 and ado-trastuzumab emtansine (T-DM1) intravenously (IV) over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity, or at the discretion of the treating physician.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed HER2-positive breast cancer that is locally advanced or metastatic (stage 4); ideally this should be from biopsy of the metastatic disease; however if this is not available, histologic confirmation from the primary tumor is acceptable
* Patients must have had progression on a trastuzumab and taxane-based chemotherapy regimen during or after treatment for locally advanced or metastatic disease or within 6 months after treatment for early-stage HER2-positive disease documented by one of the following results using Food and Drug Administration (FDA)-approved testing methods:

  * Fluorescence in situ hybridization (FISH)-positive (with an amplification ratio >= 2.0 indicating positive status) and/or
  * Immunohistochemistry (IHC) 3 + by local laboratory assessment
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must have a life expectancy >= 90 days
* Patients must have baseline laboratory tests within the following parameters at least 4 weeks (28 days) prior to registration:

  * Hemoglobin > 8 g/dL (which may be reached by transfusion)
  * Platelet count >= 100 x 10^9/L (no transfusion allowed within 2 weeks)
  * Absolute neutrophil count (ANC) >= 1.5 x 10^9/L without growth factor support
  * Serum bilirubin =< 1.5 x upper limit of normal (ULN)
  * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and/or alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 2.5 x upper limit of normal (ULN) or =< 5 x ULN if liver metastases are present
  * Serum creatinine =< 1.5 x ULN or calculated or directly measured creatinine clearance (CrCl) >= 50% LLN (lower limit of normal)
  * Fasting plasma glucose (FPG) < 140 mg/dL/7.8 mmol/L
* Patients with child-bearing potential must have a negative urine pregnancy test within 7 days prior to registration
* Patients must have a baseline electrocardiogram (ECG) showing QT interval =< 460 msec within 14 days prior to registration
* Patients must provide written informed consent prior to any registration on study
* Patients must be willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Patient must be able to swallow and retain oral medication

Exclusion Criteria:

* Patients with prior sensitivity or intolerance to PI3K inhibitors are not eligible for participation
* Patients with a history of grade >= 3 hypersensitivity reaction to trastuzumab, OR grade >= 1 with the most recent trastuzumab infusion before study entry, OR continued requirement for prolonged trastuzumab infusions to prevent hypersensitivity reactions are not eligible for participation
* Patients with a history of intolerance to trastuzumab and/or adverse events related to trastuzumab that resulted in trastuzumab being permanently discontinued are not eligible for participation
* Patients who have received prior treatment with T-DM1 are not eligible for participation
* Patients who have received prior anti-cancer therapy (e.g., biologic or other targeted therapy, chemotherapy, hormonal therapy) within 2 weeks prior to registration are not eligible for participation
* Patients with central nervous system (CNS) involvement may participate if the patient meets all of the following criteria:

  * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
  * Clinically stable with respect to the CNS tumor at the time of screening
  * Not receiving steroid therapy
  * Not receiving enzyme inducing anti-epileptic medications that were started for brain metastases
* Patients who have received radiotherapy =< 4 weeks prior to registration, with the exception of palliative radiotherapy, who have not recovered from side effects of such therapy to baseline or grade =< 1 and/or from whom >= 30% of the bone marrow was irradiated are not eligible for participation
* Patients who have undergone major surgery =< 4 weeks prior to registration or who have not recovered from side effects of such procedure are not eligible for participation
* Patients with clinically significant cardiac disease or impaired cardiac function are not eligible for participation; this includes patients with:

  * Congestive heart failure (CHF) requiring treatment (New York Heart Association [NYHA] grade >= 2)
  * Left ventricular ejection fraction (LVEF) < 50% as determined by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO)
  * Uncontrolled arterial hypertension defined by blood pressure > 140/100 mm Hg at rest (average of 3 consecutive readings)
  * History or current evidence of unstable, clinically significant cardiac arrhythmias or patients that require medications with a narrow therapeutic window, atrial fibrillation and/or conduction abnormality (e.g. congenital long QT syndrome, high-grade/complete atrioventricular [AV]-blockage)
  * Acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft [CABG], coronary angioplasty, or stenting), < 3 months prior to screening
  * QT interval adjusted according to Fridericia (QTcF) > 460 msec on screening ECG
* Patients with diabetes mellitus requiring insulin treatment and/or with clinical signs or with fasting plasma glucose (FPG) >= 140 mg/dL/7.8 mmol/L, or history of documented steroid-induced diabetes mellitus are not eligible for participation
* Patients exhibiting any other condition that would, in the Investigator's judgment, preclude patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures are not eligible for participation; this might include, but is not limited to, infection/inflammation, intestinal obstruction, and/or social/psychological complications
* Patients with impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral BYL719 (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection) are not eligible for participation
* Patients who are currently receiving medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (TdP) AND are unable to discontinue this medication or switch to a different medication prior to beginning study treatment are not eligible for participation
* Patients with a history of another malignancy within 2 years prior to registration are not eligible for participation; NOTE: the exceptions to this include cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
* Patients receiving therapeutic doses of warfarin are not eligible for participation; NOTE: Patients with a need for therapeutic anticoagulation should be given low molecular weight heparin or other non-warfarin product
* Pregnant or nursing (lactating) women are not eligible for participation; NOTE: Pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 mIU/mL)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, are not eligible for participation UNLESS they agree to use highly effective methods of contraception during dosing and for 5 weeks after study drugs discontinuation; highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject); periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least 5 weeks before receiving study treatment. In case of oophorectomy alone, the reproductive status of the woman must have been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening); for female subjects on the study the vasectomized male partner should be the sole partner for that subject
  * Combination of the following:

    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

      * NOTE: Oral contraceptives (OC), injected or implanted hormonal methods are not allowed as the sole method of contraception, as BYL719 has not been characterized with respect to its potential to interfere with the PK and/or the effectiveness of OCs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2017-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarika Jain, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on February 26, 2014 with an accrual goal of up to 28 patients. The first patient started treatment May 21 2014. The study was designed as a 3 + 3 escalation. 6 patients were enrolled in Cohort 1 and 11 patients enrolled in Cohort -1. The study closed February 12, 2016 with accrual for the study design having been met.
Groups:
- Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1): Patients receive 250 mg PO daily PI3K inhibitor BYL719 on days 1-21 and 3.6mg/kg IV over 30-90 minutes on day 1 ado-trastuzumab emtansine (T-DM1). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  PI3K inhibitor BYL719: Given PO
  Ado-trastuzumab emtansine: Given IV
  Pharmacological study: Correlative studies
  Laboratory biomarker analysis: Optional correlative studies
- Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1): Patients receive 300 mg PO daily PI3K inhibitor BYL719 on days 1-21 and 3.6mg/kg IV over 30-90 minutes on day 1 ado-trastuzumab emtansine (T-DM1). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  PI3K inhibitor BYL719: Given PO
  Ado-trastuzumab emtansine: Given IV
  Pharmacological study: Correlative studies
  Laboratory biomarker analysis: Optional correlative studies
- Cohort 2 (350mg BYL719, 3.6mg/kg T-DM1): Patients receive 350 mg PO daily PI3K inhibitor BYL719 on days 1-21 and 3.6mg/kg IV over 30-90 minutes on day 1 ado-trastuzumab emtansine (T-DM1). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  PI3K inhibitor BYL719: Given PO
  Ado-trastuzumab emtansine: Given IV
  Pharmacological study: Correlative studies
  Laboratory biomarker analysis: Optional correlative studies
- Cohort 3 (400mg BYL719, 3.6mg/kg T-DM1): Patients receive 400 mg PO daily PI3K inhibitor BYL719 on days 1-21 and 3.6mg/kg IV over 30-90 minutes on day 1 ado-trastuzumab emtansine (T-DM1). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  PI3K inhibitor BYL719: Given PO
  Ado-trastuzumab emtansine: Given IV
  Pharmacological study: Correlative studies
  Laboratory biomarker analysis: Optional correlative studies
Period: Completed 1st Cycle and Started Cycle 2
Arm/Group | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1) | Cohort 2 (350mg BYL719, 3.6mg/kg T-DM1) | Cohort 3 (400mg BYL719, 3.6mg/kg T-DM1)
Started | 11 | 6 | 0 (Due to safety data, dose was de-escalated and no patients enrolled at this dose.) | 0 (Due to safety data, dose was de-escalated and no patients enrolled at this dose.)
Completed 1st Cycle | 11 | 5 | 0 | 0
Continued on to Cycle 2 | 10 | 4 | 0 | 0
Completed | 10 | 4 | 0 | 0
Not Completed | 1 | 2 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 0
Not completed — Patient Non Compliance | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Completed 3 Cycles/Reached 1st Response
Arm/Group | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1) | Cohort 2 (350mg BYL719, 3.6mg/kg T-DM1) | Cohort 3 (400mg BYL719, 3.6mg/kg T-DM1)
Started | 10 | 4 | 0 | 0
Completed 3 Cycles | 10 | 4 | 0 | 0
Continued to Cycle 4 | 9 | 3 | 0 | 0
Completed | 9 | 3 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Progressive Disease | 1 | 1 | 0 | 0
Period: Follow Up
Arm/Group | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1) | Cohort 2 (350mg BYL719, 3.6mg/kg T-DM1) | Cohort 3 (400mg BYL719, 3.6mg/kg T-DM1)
Started | 11 | 6 | 0 | 0
Completed | 4 | 3 | 0 | 0
Not Completed | 7 | 3 | 0 | 0
Not completed — Death | 4 | 3 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- BYL719 and T-DM1 Treatment: Patients receive either 250 mg (Cohort -1) or 300 mg (Cohort 1) PO daily PI3K inhibitor BYL719 on days 1-21 and 3.6mg/kg IV over 30-90 minutes on day 1 ado-trastuzumab emtansine (T-DM1). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  PI3K inhibitor BYL719: Given PO
  Ado-trastuzumab emtansine: Given IV
  Pharmacological study: Correlative studies
  Laboratory biomarker analysis: Optional correlative studies
Arm/Group | BYL719 and T-DM1 Treatment
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
T-DM1 Systemic Therapy in Metastatic Setting [Count of Participants; unit: Participants]
  Patients had prior T-DM1 therapy | 10
  Patients had not had prior TDM1 therapy | 7
Hormone Receptor Status [Count of Participants; unit: Participants]
  Positive | 8
  Negative | 9

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) of Dose-escalating BYL719 in Combination With T-DM1
Description: DLTs of BYL719 in combination with T-DM1 will be assessed using National Cancer Institute's Common Toxicity Criteria for adverse events version 4.0 (except for hyperglycemia). A DLT is described any grade 3 or higher, clinically significant toxicity (excluding alopecia) experienced during the first 21 days following first dose of BYL719 that is determined to be at least possibly related to study medication. Lower grades may also be considered DLTs if they lead to a dose interruption of more than 7 consecutive days of BYL719. In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: The 1st 21 days (Cycle 1) of treatment
Population: 5 patients enrolled into Cohort 1 were assess for DLTs, one patient in Cohort 1 was determined not to be evaluable after review; the patient only received one dose of treatment total. Only the first 3 patients in Cohort -1 were assessed for DLTs due to 3+3 design.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1)
Number analyzed (Participants) | 3 | 5
Participants
  Thrombocytopenia | 0 | 1
  Rash Maculopapular | 0 | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD) of BYL719 in Combination With T-DM1.
Description: Safety of BYL719 in combination with T-DM1 will be assessed during the first 21 days (1 cycle=21 days) which will assist in providing the MTD. Adverse Events including dose limiting toxicities (DLT), changes in physical findings, or clinical laboratory results as well as cardiac toxicity (changes in cardiac function, which will be measured by use of echocardiogram or MUGA scan) will be evaluated.
  For each dose level, 3 patients will be treated. If none (0 of 3) show a DLT, dose will be escalated for the next cohort of patients.
  If 2 or 3 have a DLT, then the previous dose will be considered the MTD. If 2 or 3 in cohort 1 (starting dose) experience a DLT, then the dose in -1 cohort will be used.
  If 1 of 3 patients has a DLT, then an additional 3 patients will be added to that dose level.
  If 1 of 6 has a DLT, then the dose will be escalated. If 2 of 6 have a DLT, then this dose will be considered the MTD. If 3 or more of 6 have a DLT, then the previous dose will be the MTD.
Time Frame: The 1st 21 days (Cycle 1) of treatment
Population: 5 patients enrolled into Cohort 1 were assess for DLTs, one patient in Cohort 1 was determined not to be evaluable after review; the patient only received one dose of treatment total. Only the first 3 patients in Cohort -1 were assessed for DLTs due to 3+3 design in assessing for DLTs and determining the MTD.
Measure: Number; unit: mg per day
Groups:
- 250mg or 300mg BYL719, 3.6mg/kg T-DM1: Patients receive 250 mg PO daily PI3K inhibitor BYL719 on days 1-21 in Cohort -1 and 300 mg PO daily PI3K inhibitor BYL719 on days 1-21 in Cohort 1
  All patients also received 3.6mg/kg IV over 30-90 minutes on day 1 ado-trastuzumab emtansine (T-DM1). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  PI3K inhibitor BYL719: Given PO
  Ado-trastuzumab emtansine: Given IV
  Pharmacological study: Correlative studies
  Laboratory biomarker analysis: Optional correlative studies
Arm/Group | 250mg or 300mg BYL719, 3.6mg/kg T-DM1
Number analyzed (Participants) | 8
mg per day | 250

3. Secondary Outcome: Pharmacokinetics (PK) of BYL719 Administered in Combination With T-DM1.
Description: To assess the pharmacokinetics (PK)of BYL719, blood will be drawn from patients on Day 1, 8, and 15 of Cycles 1, 2 and 3 where 1 Cycle = 21 days. After that blood will be drawn once every 3 cycles. PK parameters of BYL719 including peak and trough concentrations as an estimate of the steady-state concentration, elimination clearance, interindividual variability of the elimination clearance, and the effect of PK parameters with prolonged administration of BYL719 will be obtained. Steady state concentration will be analyzed to see if there is any relationship with efficacy or toxicity.
Time Frame: Day 1, 8, and 15 of Cycles 1, 2, and 3, then every 3 Cycles (1 Cycle =21 days) while on treatment where the median number of cycles is 11 and range is 3-19 cycles.
Population: No data from the blood draws was collected or analyzed for this objective.
Arm/Group | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression-Free Survival (PFS) of BYL719 Administered in Combination With T-DM1 for All Patients Treated on Study.
Description: Progression-Free Survival (PFS) for patients treated with BYL719 and T-DM1 in combination is measured for all patients from the time of treatment initiation until the first documentation of progressive disease or death from any cause. It will be assessed every 3 months up to 1 year after discontinuation of the study drugs. Patients that completed at least 3 cycles of treatment and had imaging at 1st response time point were considered evaluable for this objective.
Time Frame: From the start of treatment and every 3 months up to 1 year after discontinuation of treatment. 1 Cycle = 21 days. Median number of cycles is 11 and range is 3-19 cycles.
Population: The sample size was so small for each cohort that it was decided that there wouldn't any merit to separating out the dose cohorts and Kaplan Meier curves were completed on all patients combined and patients with or without prior T-DM1 treatment. No data was collected and no analysis was completed on each dose cohort separately.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BYL719 and T-DM1 Treatment
Number analyzed (Participants) | 14
Months
  All Patients | 8.1 [3.9 to 10.8]
  Patients without Prior TDM1 Exposure: number analyzed (Participants) | 4
  Patients without Prior TDM1 Exposure | 10.8 [8.1 to 12.5]
  Patients with Prior TDM1 Exposure: number analyzed (Participants) | 10
  Patients with Prior TDM1 Exposure | 6.2 [1.6 to 10.5]

5. Secondary Outcome: Objective Response Rate (ORR) of BYL719 Administered in Combination With T-DM1 by Cohort
Description: ORR for patients treated with BYL719 in combination with T-DM1 assessed every 3 cycles (every 9 weeks) with imaging and Best Response defined by RECIST v1.1. ORR is defined as number of patients with Complete Response (CR)+Partial Response (PR) documented as their Best Response (confirmed 4 weeks later). Response is based on evaluation of target and non-target lesions. Clinical lesions will only be considered measurable when they are superficial. Patients that completed at least 3 cycles of treatment and had imaging at 1st response time point were considered evaluable for this objective.
  Target Lesions:
  CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of LD.
  For Non-Target Lesions:
  CR: Disappearance of all non-target lesions and normalization of tumor marker level Non-complete Response (Non-CR): Persistence of one or more non-target lesion(s)
Time Frame: From the start of treatment and every 3 cycles during treatment where 1 cycle =21 days, median number of cycles is 11 and range of cycles is 3-19.
Measure: Number; unit: participants
Arm/Group | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1)
Number analyzed (Participants) | 10 | 4
participants | 4 | 2

6. Other Pre Specified Outcome: Number of Patients With Changes in PIK3CA Gene, PTEN Expression and Akt/mTOR Downstream Markers
Description: Patients tumor tissue collected during biopsy will be evaluated by immunohitochemistry (IHC) and Next Generation Sequencing (NGS) to see if the study drugs are efficacious on patients who have this alteration.
Time Frame: Baseline
Population: The sample size was so small for each cohort and due to the exploratory nature of outcome measure, there wouldn't any merit to separating out dose cohorts. Mutations were collected for patients combined, reported on and correlated with response descriptively. No data was collected/no analysis was completed on each dose cohort separately.
Measure: Count of Participants; unit: Participants
Arm/Group | 250mg or 300mg BYL719, 3.6mg/kg T-DM1
Number analyzed (Participants) | 11
Participants
  PTEN Loss (IHC): number analyzed (Participants) | 7
  PTEN Loss (IHC) | 2
  AKT Increased Expression (IHC) | 3
  PIK3CA Mutation (NGS): number analyzed (Participants) | 6
  PIK3CA Mutation (NGS) | 4
  PI3K Pathway Aberration | 9
  Patients with Response and PTEN Loss: number analyzed (Participants) | 2
  Patients with Response and PTEN Loss | 1
  Patient with Response and AKT Increased Expression: number analyzed (Participants) | 2
  Patient with Response and AKT Increased Expression | 1
  Patient with Response and P13K Pathway Aberration: number analyzed (Participants) | 2
  Patient with Response and P13K Pathway Aberration | 2
  Patients with SD and PTEN Loss: number analyzed (Participants) | 3
  Patients with SD and PTEN Loss | 1
  Patient with SD and AKT Increased Expression: number analyzed (Participants) | 3
  Patient with SD and AKT Increased Expression | 1
  Patients with SD and PIK3CA Mutation: number analyzed (Participants) | 2
  Patients with SD and PIK3CA Mutation | 1
  Patients with SD and P13K Pathway Aberration: number analyzed (Participants) | 6
  Patients with SD and P13K Pathway Aberration | 5
  Patients with PD and PTEN Loss: number analyzed (Participants) | 1
  Patients with PD and PTEN Loss | 0
  Patients with PD and AKT Increased Expression: number analyzed (Participants) | 1
  Patients with PD and AKT Increased Expression | 0
  Patients with PD and PIK3CA Mutation: number analyzed (Participants) | 1
  Patients with PD and PIK3CA Mutation | 1
  Patients with PD and P13K Pathway Aberration: number analyzed (Participants) | 2
  Patients with PD and P13K Pathway Aberration | 1

7. Other Pre Specified Outcome: Clinical Benefit Rate (CBR) of BYL719 Administered in Combination With T-DM1 by Cohort
Description: Clinical Benefit Rate (CBR) patients treated BYL719 and T-DM1 combination treatment is defined as the number of patients with Complete Response + Partial Response + Stable Disease for over 6 months documented as their best response, assessed every 3 cycles (every 9 weeks) with physical exam and imaging (CT chest/abdomen/pelvis and bone scan, or PET/CT) and defined by RECIST guidelines. Patients that completed at least 3 cycles of treatment and had imaging at 1st response time point were considered evaluable for this objective.
Time Frame: From the start of treatment and every 3 cycles (1 cycle =21 days) while on treatment where the median number of cycles is 11 and range is 3-19 cycles.
Measure: Number; unit: participants
Arm/Group | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1)
Number analyzed (Participants) | 10 | 4
participants | 7 | 3

8. Other Pre Specified Outcome: Best Response of BYL719 Administered in Combination With T-DM1 by Cohort
Description: Best Response (BR) of patients treated with BYL719 and T-DM1 combination treatment is assessed every 9 weeks with physical exam and imaging and defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). BR is based on evaluation of target and non-target lesions. Clinical lesions will only be considered measurable when they are superficial. Patients that completed at least 3 cycles of treatment and had imaging at 1st response time point were considered evaluable for this objective.
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): >=30% decrease in the sum of the longest diameter (LD) of target lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum of LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1)
Number analyzed (Participants) | 10 | 4
participants
  Complete Response | 0 | 1
  Partial Response | 4 | 1
  Stable Disease | 5 | 1
  Progressive Disease | 1 | 1

9. Post Hoc Outcome: Toxicity of the Combination of BYL719 and T-DM1 Treatment by Cohort
Description: Toxicity profile of BYL719 in combination with T-DM1 will be assessed using National Cancer Institute's Common Toxicity Criteria for Adverse Events version 4.0 (CTCAEv4.0). Toxicity is defined as an AE that is determined to be at least possibly related to at least one of the study drugs: BYL719 and T-DM1.
  In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: From the time of treatment initiation thoughout treatment until 30 days post last dose. Range of cycles completed =1 to 19 where 1 cycle =21 days
Population: Any patient that received a dose of study drug was evaluable for this outcome measure
Measure: Number; unit: participants
Arm/Group | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1)
Number analyzed (Participants) | 11 | 6
participants
  Anemia | 0 | 1
  Pancreatitis | 0 | 1
  Electrocardiogram QT corrected interval prolonged | 0 | 1
  Lymphocyte Count Decreased | 0 | 1
  Platelet Count Decreased | 1 | 2
  Weight Loss | 1 | 0
  Anorexia | 2 | 0
  Hyperglycemia | 2 | 2
  Abnormal Uterine Bleeding | 0 | 1
  Rash Maculo-papular | 3 | 4
  Hypertension | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over 2 and half year period for all patients. Each patient was followed from the time of consent, during treatment at the beginning of each cycle through 30 days post last treatment, where 1 Cycle = 21 days the range of cycles attempted was 1-19.
Arm/Group | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1)
All-Cause Mortality (participants affected / at risk) | 4/11 | 3/6
Serious Adverse Events (participants affected / at risk) | 3/11 | 3/6
Other Adverse Events (participants affected / at risk) | 11/11 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) (N=11) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1) (N=6)
Death due to Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute pancreatitis (Gastrointestinal disorders) | 1 | 0 — Patient also experienced ascites during this SAE
Elevated Fasting Plasma (Metabolism and nutrition disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort -1 (250mg BYL719, 3.6mg/kg T-DM1) (N=11) | Cohort 1 (300mg BYL719, 3.6mg/kg T-DM1) (N=6)
Anemia (Blood and lymphatic system disorders) | 8 | 4
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 5 | 2
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Blurred Vision (Eye disorders) | 3 | 1
Dry Eye (Eye disorders) | 1 | 0
Floaters (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 3
Dry Mouth (Gastrointestinal disorders) | 4 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 5
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Chills (Gastrointestinal disorders) | 1 | 0
Edema Limbs (General disorders) | 2 | 1
Fatigue (General disorders) | 8 | 5
Fever (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Pain (General disorders) | 2 | 2
Breast Infection (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Mucosal Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 0
Wound Infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Radiation Recall Reaction (Dermatologic) (Injury, poisoning and procedural complications) | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2 | 1
Alanine Aminotransferase Increased (Investigations) | 5 | 2
Alkaline Phosphatase Increased (Investigations) | 7 | 4
Aspartate Aminotransferase Increased (Investigations) | 10 | 5
Blood Bilirubin Increased (Investigations) | 5 | 0
Creatinine Increased (Investigations) | 0 | 1
Electrocardiogram QT Corrected Interval Prolonged (Investigations) | 2 | 1
Lymphocyte Count Decrease (Investigations) | 6 | 5
Lymphocyte Count Increase (Investigations) | 1 | 0
Neutrophil Count Decrease (Investigations) | 3 | 2
Platelet Count Decrease (Investigations) | 6 | 3
Weight Loss (Investigations) | 2 | 2
White Blood Cell Decrease (Investigations) | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 7 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 4 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 9 | 2
Sinus Pain (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 3
Hypertension (Vascular disorders) | 2 | 2
Lymphedema (Vascular disorders) | 1 | 2
Nonspecific T Wave Abnormality on ECG (Cardiac disorders) | 0 | 1
Right Bundle Block (Cardiac disorders) | 1 | 0
Pancreatic Insufficiency (General disorders) | 1 | 0
Elevated Hemoglobin A1C (Investigations) | 4 | 0
Fractured Rib (Musculoskeletal and connective tissue disorders) | 1 | 0
Sebaceous Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Post- Menopausal Bleeding (Reproductive system and breast disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorder NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes